CLINICAL TRIAL: NCT05318898
Title: Effect of Dietary Protein on the Regulation of Exosome microRNA Expression in Patients
Brief Title: Effect of Dietary Protein on the Regulation of Exosome microRNA Expression in Patients With Insulin Resistance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Martha Guevara Cruz, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3986-22-22-1
Record Dates: First submitted 2022-03-24; First posted 2022-04-08 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — GDF1 protein, Xenopus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person performing the analysis of the study results should be unaware of the assigned intervention so that such knowledge does not influence the results. Therefore, it will be a person outside the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular diet with vegetable protein (Experimental): Nutritional recommendations will be given to ensure that the patient consumes a regular diet where the protein intake will be mostly from vegetable protein sources.
  Interventions: Other: Vegetal protein
- Regular diet with animal protein (Active Comparator): Nutritional recommendations will be given to ensure that the patient consumes a regular diet where the protein intake will be mostly from animal protein sources.
  Interventions: Other: Animal protein

INTERVENTIONS:
Other: Vegetal protein — Nutritional recommendations will be given to ensure that the patient consumes a regular diet where the protein intake will be mostly from vegetal protein sources
  Arms: Regular diet with vegetable protein
Other: Animal protein — Nutritional recommendations will be given to ensure that the patient consumes a regular diet where the protein intake will be mostly from animal protein sources.
  Arms: Regular diet with animal protein

SUMMARY:
miRNAs are small non-coding RNAs of approximately 22 nucleotides in length, which have the function of regulating gene expression at the post-transcriptional level through base complementation of protein-coding transcripts, this interaction leading to translational repression by destabilizing the messenger RNA. Evidence demonstrates an association between differences in miRNA expression and the development of various pathologies, including obesity, type 2 diabetes, cardiovascular disease, neurodegenerative disorders and cancer. Other factors that could also modulate miRNA expression include nutritional status, diet and even exercise. The aim of this study is to identify exosome microRNAs that modify their expression in plasma from patients with insulin resistance fed different dietary protein sources. A randomized controlled clinical trial will be performed where the selected participants will be assigned by lottery to a dietary intervention of usual diet with protein of plant or animal origin for 4 weeks. The study will consist of 3 visits where anthropometric parameters, body composition, systolic and diastolic blood pressure, dietary compliance through 24-hour recall and food logs, biochemical tests (insulin, glucose, triglycerides, total cholesterol, HDL, LDL), the relative expression of plasma exosome miRNAs and markers of oxidative stress will be evaluated. Participants will receive a weekly food pantry during the first two visits in order to improve compliance to the dietary intervention.

DETAILED DESCRIPTION:
The study will evaluate the effect of 2 dietary interventions on the regulation of plasma exosome microRNA expression in patients with insulin resistance.

STUDY PROGRAM

The study will consist of 3 visits

Planned (selection of participants)

1. Participants will be invited through advertisements.
2. Participants will be corroborated to ensure that they meet the criteria for selection.
3. If they are candidates for the protocol, participants will be provided with the letter of consent to read carefully and any doubts that may arise will be resolved. Participants will be informed about the characteristics of the study as well as the expected risks and benefits. If they agree, the participant will be asked to sign the consent form.
4. Anthropometric measurements such as weight, height, blood pressure and body composition will be determined by means of bioelectrical impedance.
5. A 24-hour reminder of food consumption will be made.
6. A whole blood sample will be taken for glucose and insulin determination, in order to determine the HOMA-Insulin Resistance index.

Once the insulin resistance patients are identified (HOMA- Insulin Resistance ≥ 2.5) the study will begin and participants will be randomized into two intervention groups.

Visit 1 (baseline)

1. A medical and nutritional assessment will be performed.
2. The physical activity questionnaire (IPAQ long version) will be administered and participants will be advised not to change their physical activity.
3. Anthropometric and blood pressure measurements will be taken.
4. Oral glucose tolerance test will be performed for 2 hours after a 12-hour fast to determine the area under the insulin and glucose curve and determination of insulinemic and glycemic indices.
5. A blood sample will be obtained to determine plasma exosome microRNA expression and C-reactive protein as a confounding variable for concurrent infection.
6. The patient will be assigned to an intervention group (vegetable protein vs. animal protein) by block randomization.
7. The participants will continue their usual diet, And the consumption of animal protein or the consumption of vegetable protein will be recommended, according to the assigned group. They will be given and explained a list of foods that provide proteins of animal and vegetable origin, which they could integrate into their usual diet, these lists will indicate which foods to consume and which not to consume, according to the intervention group to which they were assigned.

9. They will be given a logbook to write down their daily food consumption and they will be taught how to fill it out.

10. An online questionnaire will be explained how to fill out every third day to detect the consumption of recommended and non-recommended foods from the list provided, according to the assigned group.

11. They will be given a pantry with foods rich in protein only (animal protein vs. vegetable protein) according to the assigned group (explained in the section on pantries).

Visit 2 (intermediate)

1. Consumption logs will be collected.
2. The weekly pantry will be delivered
3. Clarification of doubts

Visit 3 (final)

1. A medical and nutritional assessment will be performed. 2.
2. The physical activity questionnaire (IPAQ long version) will be completed.
3. Anthropometric and blood pressure measurements will be performed.
4. Oral glucose tolerance test will be performed for 2 hours after a 12 hour fast to determine the area under the insulin and glucose curve and determination of insulinemic and glycemic indices.
5. A blood sample will be obtained to determine plasma exosome microRNA expression and C-reactive protein as a confounding variable for concurrent infection.
6. Body temperature will be determined and if female, the date of last menstrual period will be questioned as a confounding variable.
7. The food log will be collected.
8. Clarification of doubts and thanks will be given for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) between the ages of 18 and 60.
* Patients with obesity (BMI ≥ 30 and ≤ 50 kg / m2) and with insulin resistance (HOMA - Insulin Resistance Index ≥ 2.5).
* Signature of letter of consent

Exclusion Criteria:

* Patients with any type of diabetes.
* Patients with kidney disease diagnosed by a medical or with creatinine> 1.3 mg / dL for men and > 1.1 mg / dL for women and / or blood urea nitrogen > 20 mg / dL.
* Patients with acquired diseases that produce obesity and diabetes secondarily.
* Patients who have suffered a cardiovascular event.
* Patients with weight loss > 3 kg in the last 3 months.
* Patients with any catabolic diseases.
* Gravidity status
* Positive smoking and alcoholism
* Treatment with any medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in the expression profile of microRNAs from exosomes with real -time quantitative polymerase chain reaction in fold change | 4 weeks
  Fold change in the expression profile of microRNAs from exosomes after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) with real -time quantitative polymerase chain reaction

SECONDARY OUTCOMES:
Change on HOMA index | 4 weeks
  Change in the HOMA index after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal).
Change in body weight in kg | 4 weeks
  Change in the body weight in kg after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) using a standard calibrated electronic balance.
Change in biochemical parameters in mg/dL | 4 weeks
  Change the biochemical parameters in mg/dL ( glucose, total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol) after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) analysed by an enzymatic colorimetric method using the Cobas C111 analyser (Roche Diagnostic. Indianapolis. IN).
Change in body composition in percentage | 4 weeks
  Change in the body composition in percentage after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) by multifrequency bioimpedance analysis.
Change in C Reactive Protein in mg/L | 4 weeks
  Change in C Reactive Protein in mg/L after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) analysed by an enzymatic colorimetric method using the Cobas C111 analyser (Roche Diagnostic. Indianapolis. IN).
Amino acid profile in mmol/L | 4 weeks
  Change in amino acid profile in mmol/L after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) determinated by High performance liquid chromatography
Change in the area under curve of glucose in mg/dL per 2 hours | 4 weeks
  Change in the area under curve of glucose in mg/dL per 2 hours after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal).
Change in the area under curve of insulin in microIU/mL per 2 hours | 4 weeks
  Change in the area under curve of insulin in micro IU/mL per 2 hours after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal).
Change in the waist circumference in centimeters | 4 weeks
  Change in the waist circumference in centimeters after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) using a flexible tape measure.
Change in the blood pressure in mmHg | 4 weeks
  Change in the blood pressure in mmHg after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal).
Change in the Malondialdehyde in micromol/L | 4 weeks
  Change in the Malondialdehyde in micromol/L after 4 weeks of usual diet with consumption of different protein sources (vegetable vs. animal) measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Martha Guevara-Cruz, Doctor, Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran
Locations (2):
- Mexico (2):
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City
  - Martha Guevara Cruz, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lasser C. Mapping Extracellular RNA Sheds Lights on Distinct Carriers. Cell. 2019 Apr 4;177(2):228-230. doi: 10.1016/j.cell.2019.03.027. PMID 30951666
- [Background] Mori MA, Ludwig RG, Garcia-Martin R, Brandao BB, Kahn CR. Extracellular miRNAs: From Biomarkers to Mediators of Physiology and Disease. Cell Metab. 2019 Oct 1;30(4):656-673. doi: 10.1016/j.cmet.2019.07.011. Epub 2019 Aug 22. PMID 31447320
- [Background] Safdar A, Tarnopolsky MA. Exosomes as Mediators of the Systemic Adaptations to Endurance Exercise. Cold Spring Harb Perspect Med. 2018 Mar 1;8(3):a029827. doi: 10.1101/cshperspect.a029827. PMID 28490541
- [Background] Huang Y, Yan Y, Xv W, Qian G, Li C, Zou H, Li Y. A New Insight into the Roles of MiRNAs in Metabolic Syndrome. Biomed Res Int. 2018 Dec 17;2018:7372636. doi: 10.1155/2018/7372636. eCollection 2018. PMID 30648107
- [Background] Castano C, Kalko S, Novials A, Parrizas M. Obesity-associated exosomal miRNAs modulate glucose and lipid metabolism in mice. Proc Natl Acad Sci U S A. 2018 Nov 27;115(48):12158-12163. doi: 10.1073/pnas.1808855115. Epub 2018 Nov 14. PMID 30429322
- [Background] Jimenez-Lucena R, Alcala-Diaz JF, Roncero-Ramos I, Lopez-Moreno J, Camargo A, Gomez-Delgado F, Quintana-Navarro GM, Vals-Delgado C, Rodriguez-Cantalejo F, Luque RM, Delgado-Lista J, Ordovas JM, Perez-Martinez P, Rangel-Zuniga OA, Lopez-Miranda J. MiRNAs profile as biomarkers of nutritional therapy for the prevention of type 2 diabetes mellitus: From the CORDIOPREV study. Clin Nutr. 2021 Mar;40(3):1028-1038. doi: 10.1016/j.clnu.2020.06.035. Epub 2020 Jul 15. PMID 32723508
- [Background] Min KH, Yang WM, Lee W. Saturated fatty acids-induced miR-424-5p aggravates insulin resistance via targeting insulin receptor in hepatocytes. Biochem Biophys Res Commun. 2018 Sep 10;503(3):1587-1593. doi: 10.1016/j.bbrc.2018.07.084. Epub 2018 Jul 20. PMID 30033101